CLINICAL TRIAL: NCT01104220
Title: Role of Immune System in Obesity-related Inflammation and Cardiometabolic Risk
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201102127
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Non-alcoholic Fatty Liver Disease; Metabolic Syndrome; Metabolically Abnormal Obesity; Metabolically Normal Obesity; Obesity
Keywords: NAFLD; Obesity; Metabolic syndrome
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Metabolic Syndrome; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Lean, metabolically normal (No Intervention): Subjects with body mass index 18.5 - 24.9 kg/m² and normal fasting blood glucose and oral glucose tolerance and liver fat.
- Obese, metabolically normal (No Intervention): Subjects with body mass index ≥30.0 kg/m² and normal fasting blood glucose and oral glucose tolerance and liver fat.
- Obese, metabolically abnormal (No Intervention): Subjects with body mass index ≥30.0 kg/m² and impaired fasting or oral glucose tolerance and increased liver fat.
- Obese, scheduled for bariatric surgery (Experimental): Subjects with a body mass index ≥35.0 kg/m² undergoing bariatric surgery
  Interventions: Other: Weight loss
- Obese, scheduled for gallbladder surgery (No Intervention): Subjects with a body mass index ≥35.0 kg/m² undergoing gallbladder surgery
- Lean, scheduled for inguinal hernia, hysterectomy or myomectomy surgery (No Intervention): Subjects with body mass index 18.5 - 24.9 kg/m² and normal fasting blood glucose and oral glucose tolerance and liver fat.

INTERVENTIONS:
Other: Weight loss — Bariatric surgery-induced weight loss to achieve ~20%-30% reduction in initial body weight
  Arms: Obese, scheduled for bariatric surgery

SUMMARY:
The purpose of this study is to learn more about how the body stores fat in and around organs (for example in the liver) and why this affects some people's health more than others. Understanding this may lead to better treatments for diseases such as diabetes and cardiovascular disease.

DETAILED DESCRIPTION:
The purpose of this study is to determine the specific cellular and organ system metabolic and immunologic alterations that are associated with insulin resistance and inflammation in order to identify putative mechanisms and novel bio-markers involved in the pathogenesis and progression of inflammatory and cardiometabolic diseases.

ELIGIBILITY:
Inclusion Criteria:

Lean, metabolically healthy group - Body mass index (BMI) 18.5-24.9 kg/m2, HbA1C ≤5.6%, fasting plasma glucose concentration <100 mg/dl, 2-h OGTT plasma glucose concentration <140 mg/dl and intrahepatic triglyceride (IHTG) content ≤5%.

Obese, metabolically healthy group - BMI ≥30 kg/m2, HHbA1C ≤5.6%, fasting plasma glucose concentration <100 mg/dl, 2-h OGTT plasma glucose concentration <140 mg/dl and intrahepatic triglyceride (IHTG) content ≤5%.

Obese, metabolically healthy group - BMI ≥30 kg/m2, IHTG content ≥5.6% and HbA1C ≥5.7% or fasting plasma glucose concentration ≥100 mg/dl or 2-h OGTT plasma glucose concentration ≥140 mg/dl.

Lean, scheduled for inguinal hernia, hysterectomy or myomectomy surgery - BMI 18.5-24.9 kg/m2, HbA1C ≤5.6%, fasting plasma glucose concentration <100 mg/dl, 2-h OGTT plasma glucose concentration <140 mg/dl and IHTG content ≤5%.

Obese, scheduled for bariatric and gallbladder surgery - BMI ≥35.0kg/m2

Exclusion Criteria:

* active or previous history of liver diseases other than NAFLD
* history of alcohol abuse
* currently consuming ≥20 g alcohol/day
* severe hypertriglyceridemia (>300 mg/dL)
* smoke tobacco
* cancer diagnosis within the previous 5 years
* medications that might confound the study results
* pregnancy or lactation
* exercise >2 h/week

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2010-04 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | Baseline
  Insulin sensitivity assessed in vivo by using a hyperinsulinemic-euglycemic clamp procedure with stable isotope tracer infusion

SECONDARY OUTCOMES:
TNF-alpha | Baseline
  TNF-alpha is a marker of inflammation
Interleukin-6 (IL-6) | Baseline
  Interleukin-6 is a marker of inflammation
Liver tissue inflammation | Baseline
  Liver immune cell content
Abdominal adipose tissue inflammation | Baseline only in participants scheduled for bariatric surgery
  Subcutaneous, omental and transverse mesocolic adipose tissue
Abdominal adipose tissue inflammation | Baseline only in participants scheduled for gallbladder, inguinal hernia, hysterectomy or myomectomy surgery
  Subcutaneous and omental adipose tissue
Upper vs lower adipose tissue inflammation | Baseline (All groups)
  Immune cell content in abdominal and femoral subcutaneous adipose tissue
Exosome-mediated intercellular signaling | Baseline only in participants scheduled for bariatric surgery
  Signaling between cells and organs will be examined by isolating exosomes (small extracellular vesicles) from blood, subcutaneous, omental and transverse mesocolic adipose tissue and liver.
Exosome-mediated intercellular signaling | Baseline only in participants scheduled for gallbladder, inguinal hernia, hysterectomy or myomectomy surgery
  Signaling between cells and organs will be examined by isolating exosomes (small extracellular vesicles) from blood, subcutaneous and omental adipose tissue
Exosome-mediated intercellular signaling | Baseline only in all participants
  Signaling between cells and organs will be examined by isolating exosomes (small extracellular vesicles) from blood and abdominal and femoral subcutaneous adipose tissue.
Change in exosome-mediated intercellular signaling | Before and after 20-30% weight loss (~3-4 months) in participants scheduled for bariatric surgery
  Signaling between cells and organs will be examined by isolating exosomes (small extracellular vesicles) from blood and adipose tissue
Hepatic PNPLA3 synthesis rate | Baseline only in people scheduled for gallbladder or bariatric surgery
  Synthesis rates assessed by stable isotope techniques in the fasted vs the fed states

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Yoshino J, Patterson BW, Klein S. Adipose Tissue CTGF Expression is Associated with Adiposity and Insulin Resistance in Humans. Obesity (Silver Spring). 2019 Jun;27(6):957-962. doi: 10.1002/oby.22463. Epub 2019 Apr 19. PMID 31004409